CLINICAL TRIAL: NCT00003657
Title: High Dose Ifosfamide, Carboplatin and Etoposide With Amifostine Chemoprotection
Brief Title: High-dose ICE With Amifostine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul G. Richardson, MD, Richardson, Paul MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-068; P30CA006516 (NIH); DFCI-98068; ALZA-97-038-ii; NCI-V98-1491
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Bladder Cancer; Brain and Central Nervous System Tumors; Carcinoma of Unknown Primary; Extragonadal Germ Cell Tumor; Head and Neck Cancer; Kidney Cancer; Lung Cancer; Ovarian Cancer; Sarcoma; Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: metastatic osteosarcoma; recurrent non-small cell lung cancer; chondrosarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent osteosarcoma; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage IIIB non-small cell lung cancer; unspecified adult solid tumor, protocol specific; classic Kaposi sarcoma; immunosuppressive treatment related Kaposi sarcoma; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; extragonadal germ cell tumor; newly diagnosed carcinoma of unknown primary; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; borderline ovarian surface epithelial-stromal tumor; recurrent carcinoma of unknown primary; ovarian sarcoma; adult central nervous system germ cell tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; clear cell sarcoma of the kidney; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Central Nervous System Neoplasms; Neoplasms, Unknown Primary; Head and Neck Neoplasms; Kidney Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Sarcoma; Testicular Germ Cell Tumor; Osteosarcoma; Carcinoma, Non-Small-Cell Lung; Chondrosarcoma; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Testicular Neoplasms; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Amifostine; Carboplatin; Etoposide; etoposide phosphate; Ifosfamide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Dose ICF with Amifostine (Experimental): * Patients undergo peripheral blood stem cell transplantation (PBSC) harvest on day -8,
  * ifosfamide IV, carboplatin IV etoposide IV (ICE) by 96 hour continuous infusion on days -7 to -4.
  * Patients receive amifostine IV twice a day on days -7 to -3.
  * PBSCs are reinfused on day 0.
  * Filgrastim (G-CSF) is administered subcutaneously beginning on day 0 at least 2 hours after infusion of the stem cells and continuing until blood cell counts recover.
  * Patients are followed monthly for the first 2 months and then for survival.
  Interventions: Biological: filgrastim; Drug: Amifostine; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: Amifostine
  Other Names: Ethyol®
Drug: Carboplatin
  Other Names: Paraplatin
Drug: Etoposide
  Other Names: Toposar; VePesid; Etopophos
Drug: Ifosfamide
  Other Names: Ifex
Procedure: peripheral blood stem cell transplantation

SUMMARY:
The purpose of the study is to evaluate the combination of amifostine and high dose chemotherapy with blood stem cell support. Amifostine is a druf developed to protect normal tissues against the toxicities of chemotherapy and radiotherapy and has reduced the side effects of chemotherapy given at conventional doses.

ELIGIBILITY:
Eligibility Criteria:

* Histologically documented malignancy
* Metastatic or locally unresectable malignancy
* Patient may be responding to therapy

  * Responding Stage IIIC/IV or recurrent/refractory ovarian carcinoma (ineligible for other bone marrow or stem cell transplant protocols)
  * Relapsed germ cell carcinomas
  * Relapsed lymphomas (ineligible for other BMT or SCT protocols
  * SCLC in PR or CR
  * Sarcomas in or near complete remission after induction chemotherapy
  * Stage IIIB NSCLC responding to chemotherapy
  * Responsive bladder, head and neck carcinoma, or carcinoma of unknown primary
  * Other tumors without curative or first line therapy (not eligible for phase II or III studies)
* Aged 18 to 55 Physiologic years

  -- Performance status: PS 0-1
* Prior Treatment

  * > 1 week since surgery or RT
  * > 3 weeks since prior CT
* Informed Consent
* Required initial laboratory data:

  * White Cell Count Life ≥ 3000/ul
  * Platelet Count ≥ 100,000/ul
  * Creatinine ≤ 1.5 x normal
  * Bilirubin ≤ 1.5 x normal
  * No current metastases

    * BM Asp & Bx
    * Brain CAT
  * Creatinine Clearance ≥ 60 cc/min
  * SGOT < 2.5 x normal
* No other serious medical or psychiatric illness which would prevent informed consent or general anesthesia

  * Uncontrolled or severe cardiovascular disease including recent (< 6 months) myocardial infarction, or congestive heart failure
  * Active uncontrolled bacterial, viral, or fungal infection; or an active duodenal ulcer; until these conditions are corrected or controlled
  * Pregnancy
  * Unable to stop taking antihypertensive medication 24 hours prior to administration of Ethyol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1998-07; Primary Completion 2000-11 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Grade 2 or higher renal toxicities | 2 Months

SECONDARY OUTCOMES:
Full Pharmacokinetic profiles for ifosfamide and its metabolites MTD of ICE with amifostine | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paul G.G. Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elias AD, Richardson P, Tretyakov O, et al.: Amifostine with high dose infosfamide, carboplatin, and etoposide (ICE) with hematopoietic STEM cell support. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A197, 2000.